CLINICAL TRIAL: NCT03941015
Title: Tissue Oxygenation During Treatment of Infant Congenital Heart Defects
Status: Completed | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Jun Ma, the chief of department of anesthesiology, Beijing Anzhen Hospital
Other Study IDs: 2018009
Record Dates: First submitted 2018-11-19; First posted 2019-05-07 (Actual); Results first posted 2021-02-09 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Acute Kidney Injury; Hypoxia-Ischemia, Brain; Mesenteric Ischemia
Keywords: Near infrared spectroscopy; Acute Kidney Injury; congenital heart disease
MeSH Terms: conditions — Acute Kidney Injury; Hypoxia-Ischemia, Brain; Mesenteric Ischemia; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * urine samples
  * blood samples
  * stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with renal desaturation: Patients who underwent a decrease of SrtO2 measurement from the baseline value for more than 20% lasting for more than 60 s.
- patients without renal desaturation: Patients who didn't undergo a decrease of SrtO2 measurement from the baseline value for more than 20% lasting for more than 60 s.

SUMMARY:
Background: Acute kidney injury (AKI) is a common and serious postoperative complication in children with congenital heart disease. In this prospective cohort study, we tested the hypothesis that renal desaturation defined as a 20% decline of renal tissue oxygen saturation (SrtO2) from the baseline value is associated with AKI in infants undergoing ventricular septal defect (VSD) repair with cardiopulmonary bypass (CPB).

Methods: Infants aged 1 months to 12 months and scheduled to undergo VSD repair with CPB were eligible. SrtO2 was monitored using a tissue near-infrared spectroscopy. Renal desaturation was defined as a decrease of SrtO2 measurement from the baseline value for more than 20% lasting for more than 60 s. The primary outcome was the incidence of AKI on postoperative 1-3 days according to the Kidney Disease: Improving Global Outcomes criteria. The secondary outcomes included different stages of AKI, duration of postoperative mechanical ventilation, duration of intensive care unit (ICU) and hospital stay, renal replacement therapy (RRT), and in-hospital mortality.

DETAILED DESCRIPTION:
Using near-infrared spectroscopy (NIRS) to monitor intraoperative and postoperative tissue oxygen saturation and to investigate the correlation with postoperative complications.

Intraoperative hemodynamic parameters were monitored by Mostcare(PRAM, Vygon Health, Padua, Italy) including cardiac index, systemic vascular resistance index, stroke volume index, the maximal slope of systolic upstroke, cardiac cycle efficiency.

SrtO2 was monitored using a tissue near-infrared spectroscopy (FORE-SIGHT ELITE tissue oximeter, CASMED, Branford, Connecticut, USA; now acquired by Edwards Lifesciences, Irvine, California, USA). A biophotonic sensor was placed on the left flank at the level of T10-L2 to monitor SrtO2. The tissue oximeter generated a new SrtO2 data every 2 seconds. All these data were exported from the monitor as the end of surgery. As this is an observational study, the SrtO2 data were only used for research purpose, not for clinical decision making. The function of tissue oximeter was checked by a dedicated research personnel in the operating room. The infant was dropped from the study if the SrtO2 measurements were not available for more than 5 min during surgery. The baseline SrtO2 was defined as the median value of the 5-minute measurements which were measured following anesthesia induction and during the period when the cardiac index ≥2.5 L/min/m2. Renal desaturation was defined as a decrease of SrtO2 measurement from the baseline value for more than 20% lasting for more than 60 s.

The electronic data streams from the NIRS and other patient monitors will be collected into a study computer. Data collection will initiate at pre-induction of anesthesia in the operating room. Only the NIRS values will be blinded from clinical use. Blood samples for determining biomarkers of ischemic tissue injury will be taken at defined intervals. No other modifications to clinical practice will occur while conducting the study and the NIRS monitoring is non-invasive.

The primary outcome was the incidence of AKI within 3 days after surgery according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria. Secondary outcomes including different stages of AKI, duration of postoperative mechanical ventilation, duration of intensive care unit (ICU) and hospital stay, and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 1 year
2. Diagnosis of ventricular septal defect
3. Undergoing cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

1. refusal to participate;
2. emergent or urgent surgery;
3. weight >10 kg;
4. preoperative renal dysfunction;
5. multiple organ dysfunction;
6. chromosomal abnormalities;
7. skin condition precluding the application of near-infrared spectroscopy probe.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants aged 1 month to 12 months and scheduled to undergo ventricular septal defect repair with cardiopulmenary bypass were eligible.
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boqun Cui, MA, Principal Investigator — Anzhen hospital Beijing China
Locations (1):
- Anzhen hospital, Beijing, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang D, Ouyang C, Zhao X, Cui B, Dai F, Meng L, Ma J. Renal tissue desaturation and acute kidney injury in infant cardiac surgery: a prospective propensity score-matched cohort study. Br J Anaesth. 2021 Oct;127(4):620-628. doi: 10.1016/j.bja.2021.06.045. Epub 2021 Aug 24. PMID 34446224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2018 to August 2020, a total of 245 infants undergoing VSD repair with CPB in Beijing Anzhen Hospital, capital medical university were enrolled in this study.
Pre-assignment Details: Three patients were dropped due to missing data. The final analysis included 242 patients.
Groups:
- Renal Desaturation Group: Patients who underwent a decrease of SrtO2 measurement from the baseline value for more than 20% lasting for more than 60 s.
- Renal Eusaturation Group: Patients who didn't undergo a decrease of SrtO2 measurement from the baseline value for more than 20% lasting for more than 60 s.
Period: Overall Study
Arm/Group | Renal Desaturation Group | Renal Eusaturation Group
Started | 38 | 207
Completed | 38 | 204
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Population: A biophotonic sensor was placed on the left flank at the level of T10-L2 to monitor SrtO2. SrtO2 was measured during surgery. Infants who underwent at least 20% decrease in SrtO2 from the baseline level for at least 60 consecutive seconds were assigned to the renal desaturation group and other infants were assigned to the normal saturation group.
Groups:
- Patients Without Renal Desaturation: Patients who did't undergo a decrease of SrtO2 measurement from the baseline value for more than 20% lasting for more than 60 s.
- Total: Total of all reporting groups
Arm/Group | Patients With Renal Desaturation | Patients Without Renal Desaturation | Total
Number analyzed (Participants) | 38 | 204 | 242
Age, Continuous [Median (Inter-Quartile Range); unit: month] | 4.8 [3.1 to 7.5] | 5.0 [3.9 to 7.5] | 5.0 [3.8 to 6.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 93 | 106
  Male | 25 | 111 | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 38 | 204 | 242
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Median (Inter-Quartile Range); unit: kg] | 6.0 [4.8 to 6.9] | 5.9 [5.1 to 6.8] | 5.9 [5.1 to 6.8]
Height [Mean (Standard Deviation); unit: cm] | 64 (5) | 63 (6) | 64 (5)
Body surface area(BSA) [Mean (Standard Deviation); unit: m^2] | 0.31 (0.05) | 0.32 (0.05) | 0.31 (0.05)
ventricular septal defect size [Median (Inter-Quartile Range); unit: mm] | 9.0 [7.4 to 11.0] | 9.0 [7.0 to 11.0] | 9.0 [7.0 to 11.0]
Ejection fraction [Mean (Standard Deviation); unit: Percentage of blood] | 70.2 (5.9) | 70.7 (5.1) | 70.6 (5.2)
Left ventricular end-diastolic diameter [Mean (Standard Deviation); unit: mm] | 30.0 (4.5) | 29.9 (3.8) | 29.9 (3.9)
creatinine [Median (Inter-Quartile Range); unit: μmol/L] | 19.1 [16.8 to 21.6] | 18.6 [16.0 to 21.0] | 18.8 [16.1 to 21.0]
SrtO2 [Median (Inter-Quartile Range); unit: percentage of oxyhemoglobin] — SrtO2 was monitored using a tissue near-infrared spectroscopy oximeter. A biophotonic sensor was placed on the left flank at the level of T10-L2 to monitor SrtO2. SrtO2 was measured during surgery. The baseline SrtO2 was defined as the median value of the data recorded over a 5-minute epoch when the infant was induced and mechanically ventilated and had a cardiac index ≥2.5 L/min/m2, but before skin incision.
  percentage of oxyhemoglobin | 77 [74 to 79] | 75 [71 to 79] | 75 [72 to 79]
urea nitrogen [Mean (Standard Deviation); unit: mmol/L] | 3.3 (1.1) | 3.0 (1.3) | 3.1 (1.2)
hemoglobin [Mean (Standard Deviation); unit: g/L] | 11.5 (0.7) | 11.3 (0.8) | 11.4 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Kidney Injury
Description: AKI was diagnosed per the Kidney Disease: Improving Global Outcomes (KDIGO) criteria. Acute kidney injury was defined as an increase in serum creatinine to ≥1.5 times baseline within 3 days after surgery. Serum creatinine was recorded within one week before surgery and on postoperative days 1-3. Serum creatinine measured within one week before surgery was defined as serum creatinine baseline.
Time Frame: 3 days
Population: A total of 245 infants undergoing VSD repair with CPB were enrolled in this study. Three patients were dropped due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Renal Desaturation | Patients Without Renal Desaturation
Number analyzed (Participants) | 38 | 204
Participants | 18 | 57

2. Secondary Outcome: Duration of Mechanical Ventilation
Description: Hours of mechanical ventilation after surgery
Time Frame: up to 1440 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | Patients With Renal Desaturation | Patients Without Renal Desaturation
Number analyzed (Participants) | 38 | 204
hour | 51 [28 to 60] | 29 [27 to 51]

3. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay after surgery
Time Frame: up to 60 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Patients With Renal Desaturation | Patients Without Renal Desaturation
Number analyzed (Participants) | 38 | 204
day | 5 [3 to 7] | 4 [2 to 5]

4. Secondary Outcome: Duration of Stay in the Intensive Care Unit
Description: Duration of Stay in the intensive care unit after surgery
Time Frame: up to 60 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Patients With Renal Desaturation | Patients Without Renal Desaturation
Number analyzed (Participants) | 38 | 204
day | 13 [11 to 20] | 12 [10 to 15]

5. Secondary Outcome: Number of Participants Reaching Kidney Disease: Improving Global Outcomes (KDIGO) Stage 1
Description: KDIGO stage 1 was defined as serum creatinine increased more than 1.5 times serum creatinine baseline. Serum creatinine was recorded within one week before surgery and on postoperative days 1-3. Serum creatinine measured one week before surgery was defined as serum creatinine baseline. KDIGO stage 1 was considered as mild acute kidney injury.
Time Frame: 3 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Renal Desaturation | Patients Without Renal Desaturation
Number analyzed (Participants) | 38 | 204
Participants | 12 | 52

6. Secondary Outcome: Number of Participants Reaching Kidney Disease: Improving Global Outcomes (KDIGO) Stage 2
Description: KDIGO stage 2 was defined as serum creatinine increased more than 2 times serum creatinine baseline and less than 3 times serum creatinine baseline. Serum creatinine was recorded within one week before surgery and on postoperative days 1-3. Serum creatinine measured one week before surgery was defined as serum creatinine baseline. Acute kidney injury in KDIGO stage 2 was more serious than acute kidney injury in stage 1.
Time Frame: 3 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Renal Desaturation | Patients Without Renal Desaturation
Number analyzed (Participants) | 38 | 204
Participants | 4 | 4

7. Secondary Outcome: Number of Participants Reaching Kidney Disease: Improving Global Outcomes (KDIGO) Stage 3
Description: KDIGO stage 3 was defined as serum creatinine increased more than 3 times baseline, or dialysis requirement, or estimated GFR less than 35 mL/min/1.73m2. Serum creatinine was recorded within one week before surgery and on postoperative days 1-3. Serum creatinine measured one week before surgery was defined as serum creatinine baseline. Acute kidney injury in KDIGO stage 3 was more serious than acute kidney injury in stage 2.
Time Frame: 3 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Renal Desaturation | Patients Without Renal Desaturation
Number analyzed (Participants) | 38 | 204
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: collected until hospital discharge
Arm/Group | Patients With Renal Desaturation | Patients Without Renal Desaturation
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/204
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/204
Other Adverse Events (participants affected / at risk) | 0/38 | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT03941015/Prot_SAP_000.pdf